CLINICAL TRIAL: NCT04689607
Title: Comparison Between Mulligan Traction Straight Leg Raise Technique Versus Post Isometric Relaxation on Hamstring Tightness in Asymptomatic Patients
Brief Title: Mulligan Traction Straight Leg Raise Versus Post Isometric Relaxation on Hamstring Tightness in Asymptomatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rec/00676 maryam khalid abbasi
Record Dates: First submitted 2020-12-25; First posted 2020-12-30 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Hamstring Tightness
Keywords: hamstring tightness; post isometric relaxation; SLR

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Traction Straight Leg Raise (TSLR) (Experimental): This technique involves sustained traction applied to the limb. Patient actively does the SLR and both the therapist and the patient note the range. Therapist now grasp patient lower leg proximal to the ankle joint and raise it off the bed to a position just short of the painful range. Therapist flexes his knees and holds the clasped leg to his (therapist's) chest. When the therapist extends his knees this will effectively apply a longitudinal traction to the leg provided the bed is low enough and the therapist is tall enough. Sustain this traction and undertake a straight leg raise as far as it will go provided there is no pain.When pain free SLR with traction is given for three times.
  Interventions: Other: Mulligan Traction Straight Leg Raise (TSLR)
- Post Isometric Relaxation technique (PIR): (Active Comparator): The patient is placed in the supine position with the non-affected leg lying flat on the table. The knee of the affected leg is gently placed in extension, and the affected hip is then flexed. The calf of the patient is then placed on the shoulder of the practitioner The practitioner stands on the side of the affected leg. The hands of the practitioner are then placed over the upper leg, just proximal to the knee. The hip of the affected leg is then passively flexed until resistance is felt. The patient is instructed to gently attempt to push down on the practitioner's shoulder with the leg against the practitioner's resistance. The practitioner resists hip extension to create an isometric contraction and then, after appropriate time and breathing instructions. The patient is instructed to relax and the practitioner gently flexes the hip until the next barrier is reached. After a period of relaxation, the technique will be repeated three to four times.
  Interventions: Other: Post Isometric Relaxation technique (PIR):

INTERVENTIONS:
Other: Mulligan Traction Straight Leg Raise (TSLR) — The patient was in a supine position on a low bed and the therapist faced the limb of the patient that was to be treated. The therapist grasped the lower leg of the patient just near the ankle and raises the leg off the bed to a position just above the painful range. The therapist flexes the knees. Traction was retained as far as possible with a straight leg lift if there was no pain. The pain-free traction straight leg raise range was administered for 10 second and the procedure was repeated three times.
  Arms: Mulligan Traction Straight Leg Raise (TSLR)
Other: Post Isometric Relaxation technique (PIR): — The knee of the affected leg was extended, and the affected hip was flexed. Then the calf of the patient was placed on the shoulder of therapist. The therapist was standing on the side of the affected leg. The flexion of the hip was performed on the affected leg until resistance was felt. The patient was asked to gently push down on the therapist's shoulder with the leg. The therapist resisted hip extension to create an isometric contraction. The duration of the contraction was 10 seconds. Then the patient was instructed to relax and the therapist gently flexed the hip until the next barrier was felt. The technique was repeated three times.
  Arms: Post Isometric Relaxation technique (PIR):

SUMMARY:
1. Comparison between Mulligan traction straight leg raise (TSLR) and Post Isometric Relaxation (PIR) on hamstring, on range of motion (ROM) of knee extension and flexibility of hamstring muscle.
2. Secondary objective of the study is to compare the effectiveness of Mulligan Traction Straight Leg Raise (TSLR) and Post Isometric Relaxation (PIR) in lumber spine mobility in healthy individuals.
3. This study will also help to reduce the financial burden of society by identifying the commonly neglected hamstring tightness as one of the causes of developing low back pain and eventually affecting their health.
4. This study will provide evidence regarding prevention of low back pain as hamstring tightness is one of the risk factor for developing low back pain.

DETAILED DESCRIPTION:
Hamstring is the common muscle which undergoes adaptive shortening when compared with other group of muscles. Hamstrings refer to the three posterior thigh muscles and its action includes hip extension and knee flexion. Limited muscle extensibility is a common problem that affects various patient populations as well as healthy individuals. The ability of an individual to move smoothly depends on his flexibility, an attribute that enhances both safety and optimal physical activities. Flexibility is an important physiological component of physical fitness, and reduced flexibility can cause inefficiency in the workplace and is also a risk factor for low back pain. Muscle extensibility is an essential element of biomechanical function. Flexibility has been defined as the ability of a muscle to lengthen and allows one joint (or more than one joint in a series) to move through a range of motion and is an essential component of normal biomechanical functioning.

The flexibility of hamstring muscle is important for general and athletic population and of almost importance for health care professionals, to achieve this goal one needs to know the most effective and efficient technique to gain hamstring flexibility. Lack of hamstring muscles extensibility conditions decrease the pelvic mobility. This invariably leads to biomechanical changes in the pressure distribution of the spine and consequent spinal disorders. Therefore, poor hamstring extensibility has been associated with thoracic hyper kyphosis , spondylolysis , disc herniation changes in lumbopelvic rhythm and low back pain. Hamstring tightness is also associated with low back and lower extremity musculoskeletal disorders leading to biomechanical changes of the pelvis and low back. The literature reports a number of associated benefits of flexibility including improved athletic performance, reduced injury risk, prevention or reduction of post-exercise soreness, and improved coordination.

Stretching techniques are the treatments used to improve muscular extensibility to improve range of motion (ROM), and can help prevent damage in daily life or sports, reduce muscle pain, and improve muscle capability. There are various treatment for the hamstring stretching like active release technique, passive stretching, static stretching, Proprioceptive neuromuscular facilitation Stretching Techniques, eccentric stretching exercises for improving hamstring flexibility.

Mulligan performs mobilization procedures while patients were moving, either actively or passively, or while they were performing a resisted muscle contraction .Indications for use of Mulligan's Traction Straight Leg Raise (TSLR) technique are limited range of motion of hip flexion together with low back pain with or without referred leg pain. The intention of this technique is to restore normal mobility. It stretches the lower extremity muscles in combination of hamstring, adductors and rotators. The Traction Straight Leg Raise technique is painless intervention that is said to have immediate benefits.

Muscle energy technique (MET) is a procedure that involves voluntary contraction of a patient's muscle in a precisely controlled direction, at varying levels of intensity. It is unique in its application as the patient provides the initial effort while the practitioner facilitates the process. The benefits of muscle energy techniques (MET) include: Restoring normal tone in hypertonic muscles, strengthening weak muscles, preparing the muscle for subsequent stretching, improved joint mobility. It includes two techniques post isometric relaxation technique and reciprocal inhibition.

According to a study muscle energy technique (post isometric relaxation technique - PIR) is more effective than ultrasound therapy with active static stretching and passive static stretching in improving the hamstring flexibility in individuals with hamstring tightness.A study compared two muscle energy techniques (MET with 30-s post isometric stretch phase vs MET with 3-s post-isometric stretch phase) for increasing flexibility of the hamstring muscle group and concluded that both techniques appeared to be equally effective in increasing hamstring extensibility. The findings suggest that altering the duration of the passive stretch component does not have a significant impact on the efficacy of MET for short-term increase in muscle extensibility.

According to a study Mulligan traction straight leg raise technique is significantly effective in increasing straight leg raise (SLR) range of movement .A study demonstrated that both Mulligan traction straight leg raise (TSLR) and MET are effective in improving Knee range of motion (ROM) in subject with tight hamstring. The study showed that MET is significantly better then Mulligan traction straight leg raise (TSLR).The Effects of Hold-Relax Technique and Mulligan's Straight Leg Raise with Traction Technique on Flexibility of Shortened Hamstring was studied and concluded that both Mulligan's straight leg raise with traction technique and hold-relax technique show immediately. Although Mulligan's straight leg raise with traction technique was more increased average extension angle of knee joint at 90-90 straight leg raise test than the hold-relax technique.A study compared immediate effects of traction straight leg and bent leg raise on hamstring muscle flexibility in normal individuals and concluded that Mulligan's traction straight leg raise technique was more effective in improving hamstring flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic
* 20-70 degrees active knee extension loss with hip in 90 degrees flexion in dominant limb.

Exclusion Criteria:

* Volunteers involved in recreational or flexibility sport activities.
* History of previous lower limb injury from past one year.
* History of fracture or surgery of back, pelvis, hip or knee.
* Spinal deformity.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension test (Popliteal angle): | for two weeks
  Position the extremity which is being tested in hip 90 degrees of flexion,0 degrees of abduction, adduction, and rotation.The knee that is being tested is relaxed in flexion.The opposite limb will rest on the examining table with the knee positioned in full extension and the hip in 0 degrees of extension, flexion, adduction abduction, and rotation. Stabilize the femur to maintain the hip in 90 degrees of flexion and to avoid unnecessary movement at hip joint. Extend the knee to the end point when resistance is felt from development of tension in the posterior thigh muscles and upon further knee extension causes the hip extension. Measurement of knee ROM the landmarks are greater trochanter, lateral condyle of femur and the lateral malleolus. On lateral condyle of femur the fulcrum of the goniometer will be placed, the proximal arm fixed along the femur using greater trochanter as reference.The distal arm will be aligned with the lower leg using the lateral malleolus as reference.
Modified Modified Schober's Technique for lumber flexion: | for two weeks
  The investigator knelt behind standing patient and marked the Posterior superior iliac spine by labeling with her thumbs the inferior margins of the Posterior superior iliac spine of the subject. Along the midline of the lumbar spines horizontal to the Posterior superior iliac spine ,an ink mark was drawn.15 cm above the original mark, another ink mark was made. Between the skin markings, the tape measure was then lined up. The therapist instructed the subject to bend forward with the tape measure firmly pressed against the skin of the subject, and while holding the tape measure with his or her fingertips. The new distance between the superior and inferior skin markings was measured when the subject bent forward into complete lumbar flexion. After trunk flexion, the distance between these marks was measured and the change in the gap between the marks was used to demonstrate the amount of lumbar flexion. All skin marks were cleaned using rubbing alcohol after each measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Institute of Rehabilitation Sciences, Mānsehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith M, Fryer G. A comparison of two muscle energy techniques for increasing flexibility of the hamstring muscle group. J Bodyw Mov Ther. 2008 Oct;12(4):312-7. doi: 10.1016/j.jbmt.2008.06.011. Epub 2008 Aug 6. PMID 19083689
- [Background] Wang SS, Whitney SL, Burdett RG, Janosky JE. Lower extremity muscular flexibility in long distance runners. J Orthop Sports Phys Ther. 1993 Feb;17(2):102-7. doi: 10.2519/jospt.1993.17.2.102. PMID 8467336
- [Background] Dalyan M, Sherman A, Cardenas DD. Factors associated with contractures in acute spinal cord injury. Spinal Cord. 1998 Jun;36(6):405-8. doi: 10.1038/sj.sc.3100620. PMID 9648196
- [Background] Fisk JW, Baigent ML, Hill PD. Scheuermann's disease. Clinical and radiological survey of 17 and 18 year olds. Am J Phys Med. 1984 Feb;63(1):18-30. PMID 6230938
- [Background] Standaert CJ, Herring SA. Spondylolysis: a critical review. Br J Sports Med. 2000 Dec;34(6):415-22. doi: 10.1136/bjsm.34.6.415. PMID 11131228
- [Background] Harvey J, Tanner S. Low back pain in young athletes. A practical approach. Sports Med. 1991 Dec;12(6):394-406. doi: 10.2165/00007256-199112060-00005. PMID 1838423
- [Background] Esola MA, McClure PW, Fitzgerald GK, Siegler S. Analysis of lumbar spine and hip motion during forward bending in subjects with and without a history of low back pain. Spine (Phila Pa 1976). 1996 Jan 1;21(1):71-8. doi: 10.1097/00007632-199601010-00017. PMID 9122766
- [Background] Biering-Sorensen F. Physical measurements as risk indicators for low-back trouble over a one-year period. Spine (Phila Pa 1976). 1984 Mar;9(2):106-19. doi: 10.1097/00007632-198403000-00002. PMID 6233709
- [Background] Li Y, McClure PW, Pratt N. The effect of hamstring muscle stretching on standing posture and on lumbar and hip motions during forward bending. Phys Ther. 1996 Aug;76(8):836-45; discussion 845-9. doi: 10.1093/ptj/76.8.836. PMID 8710963
- [Background] Hartig DE, Henderson JM. Increasing hamstring flexibility decreases lower extremity overuse injuries in military basic trainees. Am J Sports Med. 1999 Mar-Apr;27(2):173-6. doi: 10.1177/03635465990270021001. PMID 10102097
- [Background] Marques AP, Vasconcelos AA, Cabral CM, Sacco IC. Effect of frequency of static stretching on flexibility, hamstring tightness and electromyographic activity. Braz J Med Biol Res. 2009 Oct;42(10):949-53. doi: 10.1590/s0100-879x2009001000012. PMID 19784479
- [Background] Malliaropoulos N, Mendiguchia J, Pehlivanidis H, Papadopoulou S, Valle X, Malliaras P, Maffulli N. Hamstring exercises for track and field athletes: injury and exercise biomechanics, and possible implications for exercise selection and primary prevention. Br J Sports Med. 2012 Sep;46(12):846-51. doi: 10.1136/bjsports-2011-090474. Epub 2012 Jun 9. PMID 22685125
- [Background] Larsen B, Andreasen E, Urfer A, Mickelson MR, Newhouse KE. Patellar taping: a radiographic examination of the medial glide technique. Am J Sports Med. 1995 Jul-Aug;23(4):465-71. doi: 10.1177/036354659502300417. PMID 7573659
- [Background] Elias LJ, Bryden MP, Bulman-Fleming MB. Footedness is a better predictor than is handedness of emotional lateralization. Neuropsychologia. 1998 Jan;36(1):37-43. doi: 10.1016/s0028-3932(97)00107-3. PMID 9533385
- [Background] Schneiders AG, Sullivan SJ, O'Malley KJ, Clarke SV, Knappstein SA, Taylor LJ. A valid and reliable clinical determination of footedness. PM R. 2010 Sep;2(9):835-41. doi: 10.1016/j.pmrj.2010.06.004. PMID 20869683
- [Background] van Melick N, Meddeler BM, Hoogeboom TJ, Nijhuis-van der Sanden MWG, van Cingel REH. How to determine leg dominance: The agreement between self-reported and observed performance in healthy adults. PLoS One. 2017 Dec 29;12(12):e0189876. doi: 10.1371/journal.pone.0189876. eCollection 2017. PMID 29287067
- [Background] Williams R, Binkley J, Bloch R, Goldsmith CH, Minuk T. Reliability of the modified-modified Schober and double inclinometer methods for measuring lumbar flexion and extension. Phys Ther. 1993 Jan;73(1):33-44. PMID 8417457